CLINICAL TRIAL: NCT03137745
Title: To Study the Changes in Coagulation Profile in Patients Undergoing CRS(CYTOREDUCTIVE SURGERY) and HIPEC(HYPERTHERMIC INTRAPERITONEAL CHEMOTHERAPY)
Brief Title: Coagulation Profile of Patients Undergoing CRS(Cytoreductive Surgery) and Hyperthermic Intraperitoneal Chemotherapy
Status: Completed | Type: Observational
Sponsor: Rajiv Gandhi Cancer Institute & Research Center, India (Other)
Responsible Party: Principal Investigator, Dr soumi pathak, Dr Soumi Pathak Principal Investigator, Rajiv Gandhi Cancer Institute & Research Center, India
Other Study IDs: RGCI ID:395/AN/FSP-08
Record Dates: First submitted 2017-04-26; First posted 2017-05-03 (Actual); Last update posted 2017-05-05 (Actual); Status verified 2017-04

CONDITIONS: Haematological Abnormality
Keywords: Thromboelastography, chemotherapy,hyperthermic
MeSH Terms: conditions — Fever | interventions — Thrombelastography

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- all patients undergoing CRS with HIPEC: thromboelastography was done in 60 patients undergoing CRS with HIPEC in RGCI FROM MARCH2015- MARCH 2016
  Interventions: Other: thromboelastography

INTERVENTIONS:
Other: thromboelastography — thromboelastography was done pre HIPEC ,post HIPEC and first and second postoperative days

SUMMARY:
To study the changes in coagulation profile in patients undergoing cytoreductive surgery and Hyperthermic intraperitoneal chemotherapy. The objective of the study is to determine the utility of thromboelastography in comparison to standard coagulation tests in assessing the coagulopathy in patients undergoing CRS with HIPEC.

DETAILED DESCRIPTION:
This is a prospective observational study conducted in 60 patients undergoing CRS with HIPEC in RGCIRC from march 2015- march2016 after taking permission from the institutional review board and informed written consent from the patients.

Arterial blood samples were collected before and after HIPEC and on first and second postoperative day for PT,APTT INR,TEG and ABG. Statistical analysis was done using chi square test and unpaired t- test for categorical and continuous variables. Pearson's correlation coefficient was calculated for analysing the correlation between the variables .P - value <0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* ASA 1&2
* Undergoing CRS with HIPEC

Exclusion Criteria:

* extremities of age
* patients with coagulopathy
* patients on anticoagulant preoperatively sever organ dysfunctions

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: thromboelastography was done in 60 patients undergoing CRS with HIPEC in RGCI FROM MARCH2015- MARCH 2016
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2015-03; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
comparison of thromboelastograph values with standard coagulation tests | 1.5 hours after HIPEC
  arterial samples were taken for thromboelastography and prothrombin time(seconds), fibrinogen( mg) and patial thromboplastin time( seconds)

SECONDARY OUTCOMES:
comparison of various thromboelastograph values with standard coagulation tests | 24hours and 48 hours after HIPEC
  arterial samples were taken for thromboelastography and prothrombin time(seconds), fibrinogen( mg) and partial thromboplastin time(seconds)

REFERENCES:
- [Background] Sheshadri DB, Chakravarthy MR. Anaesthetic Considerations in the Perioperative Management of Cytoreductive Surgery and Hyperthermic Intraperitoneal Chemotherapy. Indian J Surg Oncol. 2016 Jun;7(2):236-43. doi: 10.1007/s13193-016-0508-2. Epub 2016 Feb 20. PMID 27065715
- [Result] Korakianitis O, Daskalou T, Alevizos L, Stamou K, Mavroudis C, Iatrou C, Vogiatzaki T, Eleftheriadis S, Tentes AA. Lack of significant intraoperative coagulopathy in patients undergoing cytoreductive surgery and hyperthermic intraperitoneal chemotherapy (HIPEC) indicates that epidural anaesthesia is a safe option. Int J Hyperthermia. 2015;31(8):857-62. doi: 10.3109/02656736.2015.1075606. Epub 2015 Oct 8. PMID 26446799